CLINICAL TRIAL: NCT03897192
Title: Long-term Outcome of Punctate Inner Choroidopathy or Multifocal Choroiditis With Active Choroidal Neovascularization Managed With Anti-vascular Endothelial Growth Factor
Brief Title: Long-term Outcome of Zonal Outer Retinopathy in Punctate Inner Choroidopathy or Multifocal Choroiditis
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, San Ni Chen, Department of Ophthalmology, Changhua Christian Hospital
Other Study IDs: 190318
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Punctate Inner Choroidopathy
Keywords: punctate inner choroidopathy; multifocal choroiditis; zonal outer retinopathy; long-term outcome
MeSH Terms: conditions — White Dot Syndromes; Multifocal Choroiditis | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Bevacizumab — Anti-vascular endothelial growth factor (VEGF)

SUMMARY:
To report the long term prognosis in patients with punctate inner choroidopathy (PIC) or multifocal choroiditis (MFC) and associated zonal outer retinopathy (ZOR).

ELIGIBILITY:
Inclusion Criteria:

* Patients with punctate inner choroidopathy (PIC) or multifocal choroiditis (MFC) and associated zonal outer retinopathy (ZOR).
* Follow up over 4 years.

Exclusion Criteria:

* Patients with punctate inner choroidopathy (PIC) or multifocal choroiditis (MFC) without zonal outer retinopathy (ZOR).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We included patients of PIC/MFC and ZOR with a clinical follow up of 4 years or longer. Patients were recorded of age, sex, best corrected visual acuity (BCVA), refractive status, coexistence of choroidal neovascularization, number and total area of PIC/MFC lesions, treatment, and recurrent activity.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Wilcoxon Signed-Rank test | Baseline, 4 year
  A statistical comparison of average of different time point

SECONDARY OUTCOMES:
visual acuity | Baseline, 6 month, 12 month, 24 month, 36 month, 48 month
  visual acuity change in logMAR in different time point

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided